CLINICAL TRIAL: NCT05094999
Title: Assessment of the Effects of Early Proprioceptive Stimulations in Patients With Severe Traumatic Brain Injury : a Randomized Controlled Trial
Brief Title: Assessment of the Effects of Early Proprioceptive Stimulations in Patients With Severe Traumatic Brain Injury
Acronym: TC-Mouv
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A02583-36
Record Dates: First submitted 2021-09-22; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Traumatic Brain Injuries
Keywords: traumatic brain injuries; proprioceptive stimulation; vibration; spasticity; intensive care units
MeSH Terms: conditions — Brain Injuries, Traumatic; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the intervention group will receive proprioceptive stimulations set to create illusions of movement.
  Interventions: Device: Proprioceptive stimulations
- Control group (Sham Comparator): Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the control group will receive sham stimulations.
  Interventions: Device: Sham stimulations

INTERVENTIONS:
Device: Proprioceptive stimulations — Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the intervention group will receive proprioceptive stimulations set to create illusions of movement.
  Arms: Intervention group
Device: Sham stimulations — Vibration treatment will last eight weeks for each patient, with 4 sessions per week, 30 minutes per session. Subjects of the control group will receive sham stimulations.
  Arms: Control group

SUMMARY:
"Severe traumatic brain injury (TBI) is a serious condition, common in young adults. It leads to sensorimotor and cognitive sequelae that hinder social reintegration. Neuronal plasticity must be used quickly before natural recovery impedes neuronal regrowth. In this respect, stopping sedation as soon as possible and early mobilization, even if the patients are unconscious, are recognized as useful measures to promote recovery. However, at the early stage, the environment of the ICU and the acute condition of the patients limit the rehabilitation possibilities. In such a context, functional proprioceptive stimulations (Vibramoov™ system, Techno Concept, France) could be a tool of interest.

By using the proprioceptive signatures of cyclic movements, proprioceptive stimulations can elicit the illusion of these movements. A motor response can even be obtained through the interactions between the peripheral nervous system and the central nervous system. Finally, such stimulations facilitate the initiation of the mimicked movements. Some studies have already shown the benefits of proprioceptive vibrations. However, so far, these benefits have only been studied at the chronic stage of neurological diseases. The investigators hypothesized that early functional proprioceptive stimulations (FPS) may reduce spasticity and promote recovery in patients with severe traumatic brain injury.

To test the hypothesis, the investigators conduct a randomized controlled trial on patients with severe traumatic brain injury. Every patient will be included as soon as possible in the ICU and receive either FPS, either sham stimulations to the joints of the lower limbs, 4 times a week during 8 weeks. The primary outcome measures will assess spasticity. The investigators also assess pain, coma recovery; muscle wasting and cognitive impairments. "

ELIGIBILITY:
Inclusion Criteria:

* Severe TBI : Glasgow coma score (GCS) ≤ 8 (11)
* Age ≥ 18 years old
* No pregnancy
* Not being under guardianship
* Be affiliated to the French social security system

Exclusion Criteria:

* Orthopedic lesions or any medical condition that prevent the implementation of the protocol within ten days post-injury
* Traumatic SCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Changes in the modified Ashworth scale (MAS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The MAS enables to assess spasticity. The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (Score range from 0 to 5 per muscle, higher values represent a higher severity of spasticity) adductors and gracilis
Changes in the angles of the muscle reaction in the modified Tardieu scale (MTS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The MTS enables to assess the severity of spasticity. The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (The outcome is reported in degree, from 0 to 180 degrees, higher values represent a higher dynamic component of spasticity)
Changes in the quality of the muscle reaction in the modified Tardieu scale (MTS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  The muscle whose spasticity will be assessed are the soleus, gastrocnemius, knee extensors, knee flexors, adductors and gracilis (Score range from 0 to 5 per muscle, higher values represent a higher severity of spasticity)
Changes in the Spinal cord assessment tool for spastic reflexes (SCATS) | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  This score enables to asses global spasticity (Score range from 0 to 18, higher values represent a higher degree of spasticity)

SECONDARY OUTCOMES:
Changes in the visual analog scale for the auto-assessment of problematic spasticity | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury.
  Score range from 0 to 100, higher values represent a higher degree of problematic spasticity.
Changes in the visual analog scale for the auto-assessment of problematic spasticity | Every week during the eight weeks of treatment, then at 2 months (end of treatment), 6 months and 1 year after the injury
  Score range from 0 to 100, higher values represent a higher degree of problematic spasticity.
Changes in the Coma recovery scale-revised (CRS-R) | At inclusion, and at one month, 2 months and 1 year after the injury.
  This measure enables to assess coma recovery (Score range from 0 to 23, higher values represent a better outcome)
Changes in the Glasgow outcome scale (GOS) | At inclusion, and at one month, 2 months and 1 year after the injury.
  This measure enables to assess coma recovery (Score range from 0 to 5, higher values represent a better outcome)
Changes in the Glasgow outcome scale-extended (GOS-E) | At inclusion, and at one month, 2 months and 1 year after the injury.
  This measure enables to assess coma recovery (Score range from 0 to 8, higher values represent a better outcome)
Changes in the Disability rating scale (DRS) | At inclusion, and at one month, 2 months and 1 year after the injury.
  This measure enables to assess coma recovery (Score range from 0 to 29, lower values represent a better outcome)
Changes in the quadriceps muscle thickness | At inclusion, then once a week during the first month, and at 2 months, 6 months and 1 year after the injury
  "Measured with ultrasound, average of two measures (at the border between the lower third and upper two-thirds between the anterior superior iliac spine and the upper pole of the patella, and at the midpoint between the anterior superior iliac spine and the upper pole of the patella) (Measure in centimeters, higher values represent a better outcome)"
Changes in the Montreal cognitive assessment (MoCA) | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Score range from 0 to 30, higher values represent a better outcome)
Changes in the time to complete the bells cancellation test to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Measure in minutes and seconds, lower values represent a better outcome)
Changes in the digit span test to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Higher values represent a better outcome)
Changes in the Posttraumatic stress disorder checklist scale (PCLS) to assess cognitive impairments | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Score range from 17 to 85, lower values represent a better outcome)
Changes in the Hospital anxiety and depression scale (HAD scale) | Up to 1 month, then at 2 months and 1 year after the injury
  This measure enables to assess cognitive impairments (Score range from 0 to 42, lower values represent a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard VIGUE, Principal Investigator — APHP
Locations (1):
- Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No